CLINICAL TRIAL: NCT03022773
Title: Macular Pigment Measurements in Eye & Other Tissues
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Paul S. Bernstein, Professor, Ophthalmology/Visual Sciences, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB # 80132
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Macular Pigmentation; Skin Pigment
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carotenoid measurements (Other): Subjects are asked to have carotenoid levels measured in the eye, skin and/or blood.
  Interventions: Other: Carotenoid measurements

INTERVENTIONS:
Other: Carotenoid measurements — Carotenoid measurements of the eye (macula) are obtained through non-invasive ophthalmic photographs using the Heidelberg Spectralis imaging system.
  Carotenoid measurements of the skin are measured by a laboratory instrument that uses a painless blue laser light for exposure of the skin and a photodetector for scattered light.
  Carotenoid measurements in the blood are obtained through routine venipuncture.

SUMMARY:
The purpose of this study is to understand the role of nutrition and its effects on the eye and other tissues. The investigators propose to study this by validating and correlating various non-invasive measurement methods of carotenoid concentrations in the human eye and skin tissue.

A secondary objective is to correlate blood levels of carotenoids on a sub-set of participants.

DETAILED DESCRIPTION:
The macula of the human retina (the structure responsible for high acuity vision essential for reading, driving and recognizing faces) is colored an intense yellow due to the deposition of two carotenoid compounds, lutein and zeaxanthin. These xanthophyll carotenoids are derived exclusively from the diet, and are hypothesized to protect the macula from light-induced oxidative damage by virtue of their light-screening and antioxidant properties.

Epidemiological studies have shown that high dietary intake and blood levels of lutein and zeaxanthin are associated with lower rates of vision loss due to age-related macular degeneration (AMD).

It is of interest to correlate carotenoid levels in the eye and skin tissues with blood levels of carotenoid compounds.

ELIGIBILITY:
Inclusion Criteria:

* Any patient age 7 or older, undergoing routine dilated ophthalmology examinations at the Moran Eye Center will be eligible to participate.
* Patients with adult vitelliform dystrophy. (This condition initially presents in adulthood as bilateral subtle and often asymptomatic macular lesions, which are often misdiagnosed as early age-related macular degeneration (AMD)).

Exclusion Criteria:

* Patients under age 7 will not be eligible to participate.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Carotenoid levels in the eye | at enrollment
  all study procedures are generally completed in a single study visit
Carotenoid levels in the skin | at enrollment
  all study procedures are generally completed in a single study visit

SECONDARY OUTCOMES:
Carotenoid levels in the blood | at enrollment
  all study procedures are generally completed in a single study visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bernstein, MD, PhD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No